CLINICAL TRIAL: NCT01213511
Title: Neurocognitive Outcome After Coronary Artery Bypass Surgery Using Minimal Versus Conventional Extracorporeal Circulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AHEPA University Hospital (Other)
Responsible Party: Principal Investigator, Kyriakos Anastasiadis, Head of Cardiothoracic Department, AHEPA University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AHEPA_CTS-02
Record Dates: First submitted 2010-10-01; First posted 2010-10-04 (Estimated); Last update posted 2013-11-28 (Estimated); Status verified 2013-11

CONDITIONS: Coronary Artery Bypass
Keywords: coronary artery disease; coronary artery bypass grafting; cardiopulmonary bypass; minimal extracorporeal circulation
MeSH Terms: conditions — Coronary Artery Disease | interventions — Coronary Artery Bypass

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MECC Group (Active Comparator): Patients operated for elective coronary artery bypass grafting with the use of minimal extracorporeal circulation.
  Interventions: Procedure: Coronary artery bypass grafting with the use of minimal extracorporeal circulation
- CECC Group (Active Comparator): Group of patients undergoing elective coronary bypass grafting with the use of conventional extracorporeal circulation.
  Interventions: Procedure: Coronary artery bypass grafting under conventional extracorporeal circulation

INTERVENTIONS:
Procedure: Coronary artery bypass grafting with the use of minimal extracorporeal circulation — The MECC system (Maquet Cardiopulmonary, Hirlingen, Germany) consists of a pre-connected closed CPB circuit containing a RotaFlow centrifugal pump and a Quadrox D diffusion membrane oxygenator. A flow meter and a bubble sensor are integrated in the drive unit of the centrifugal pump. The system features a tip-to-tip heparin coating (Bioline Coating, Maquet Cardiopulmonary, Hirlingen, Germany). No arterial or venous line filters are included. Initial priming volume of the system is 500 mL, while using retrograde autologous priming (RAP) the circuit could be filled in with autologous blood, thus reducing hemodilution. Since no cardiotomy suction is used, shed blood is collected with a cell-saving device (Haemonetics Corp, Braintree, MA).
  Arms: MECC Group
Procedure: Coronary artery bypass grafting under conventional extracorporeal circulation — A standard open CPB circuit is used, consisting of uncoated PVC tubing, a hard-shell venous reservoir, a microporous membrane oxygenator (Dideco, Mirandola, Italy) and a roller pump (Stöckert S3, Munich, Germany). The circuit contains a 40 μm arterial line blood filter (Dideco, Mirandola, Italy) and it is primed with 1500 mL of a balanced crystalloid/colloid solution (1000 mL of Ringer's solution, 200 mL of mannitol 20%, and 300 mL of hydroxyethyl starch 6%). Cardiotomy as well as sump sucker are integrated to the circuit.
  Arms: CECC Group

SUMMARY:
The aim of this study is to assess the effect of minimal (MECC) versus conventional (CECC) extracorporeal circulation on neurocognitive function after elective coronary bypass grafting (CABG) as well as whether this can be attributed to improved cerebral perfusion intraoperatively.

DETAILED DESCRIPTION:
Despite improvements in the biocompatibility of cardiopulmonary bypass (CPB) circuits, the activation of inflammatory systemic response can result in clinically relevant organ dysfunction. Regarding the central nervous system, prolonged hypoperfusion and microembolization during conventional CPB have been related to postoperative neurologic impairment with an incidence varying from 30% to 60%. This clinical scenario covers a spectrum from a transient subtle cognitive dysfunction to a permanent stroke. Postoperative cognitive decline (POCD) is characterized as impairment in attention, cognition, recognition, orientation, memory, and learning. It may result in prolonged hospitalization, increased morbidity and mortality, while it has an adverse impact on quality of life after surgery.

Near-infrared spectroscopy (NIRS) provides a continuous and noninvasive monitoring of regional cerebral oxygen saturation (rSO2). Recent studies have shown a significant relationship between intraoperative cerebral oxygen desaturation, indicative of cerebral ischemia, and early POCD in patients undergoing elective coronary bypass grafting (CABG) with conventional extracorporeal circulation (CECC). In an attempt to reduce CPB-inherent side effects, a minimal extracorporeal circulation (MECC) system was developed and it is evaluated in clinical practice. The aim of this pilot study was to define whether there is a difference in early postoperative neurocognitive functioning between patients being operated for CABG on MECC versus CECC systems as well as whether this can be attributed to improved cerebral perfusion intraoperatively.

ELIGIBILITY:
Inclusion Criteria:

* All patients scheduled for elective coronary artery bypass grafting

Exclusion Criteria:

* history of psychiatric disorder
* inability to undergo neuropsychological assessment
* history of transient ischemic attack or stroke
* carotid artery stenosis > 60% assessed by duplex ultrasonography

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2009-01; Primary Completion 2011-01 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Neurocognitive outcome at 3-month follow-up | 3 months
  Neurocognitive outcome at 3-month follow-up after elective coronary artery bypass grafting with the use of minimal (MECC) versus conventional (CECC) extracorporeal circulation.

SECONDARY OUTCOMES:
Neurocognitive outcome at discharge | 7-30 days
  Neurocognitive score assessed at the time of discharge after elective coronary surgery with the use of minimal (MECC) versus conventional (CECC) extracorporeal circulation.
Episodes of intraoperative cerebral desaturation | During the operation
  Number of episodes and duration of cerebral desaturation assessed with the use of near-infrared spectroscopy after elective coronary artery bypass grafting with minimal (MECC) versus conventional (CECC) extracorporeal circulation.

CONTACTS AND LOCATIONS:
Overall Officials: Kyriakos Anastasiadis, FETCS, Principal Investigator — Department of Cardiothoracic Surgery, AHEPA University Hospital, Thessaloniki, Greece; Christos Papakonstantinou, Professor, Study Chair — Department of Cardiothoracic Surgery, AHEPA University Hospital, Thessaloniki, Greece
Locations (1):
- Department of Cardiothoracic Surgery, AHEPA University Hospital, Thessaloniki, Greece

REFERENCES:
- [Background] Murkin JM, Newman SP, Stump DA, Blumenthal JA. Statement of consensus on assessment of neurobehavioral outcomes after cardiac surgery. Ann Thorac Surg. 1995 May;59(5):1289-95. doi: 10.1016/0003-4975(95)00106-u. No abstract available. PMID 7733754
- [Background] Liebold A, Khosravi A, Westphal B, Skrabal C, Choi YH, Stamm C, Kaminski A, Alms A, Birken T, Zurakowski D, Steinhoff G. Effect of closed minimized cardiopulmonary bypass on cerebral tissue oxygenation and microembolization. J Thorac Cardiovasc Surg. 2006 Feb;131(2):268-76. doi: 10.1016/j.jtcvs.2005.09.023. Epub 2006 Jan 18. PMID 16434253
- [Derived] Anastasiadis K, Argiriadou H, Kosmidis MH, Megari K, Antonitsis P, Thomaidou E, Aretouli E, Papakonstantinou C. Neurocognitive outcome after coronary artery bypass surgery using minimal versus conventional extracorporeal circulation: a randomised controlled pilot study. Heart. 2011 Jul;97(13):1082-8. doi: 10.1136/hrt.2010.218610. Epub 2011 Feb 28. PMID 21357641
- See also: CardioThoracic Surgery Network — http://www.ctsnet.org